CLINICAL TRIAL: NCT07270874
Title: LIVER AKI: A Randomized, Open-label Trial to Evaluate the Efficacy of Intravenous Human Albumin Administration Versus Saline Solution (NaCl 0.9%) in Patients With descompénsate Cirrhosis and AKI 1B or Grater
Brief Title: Study to Evaluate the Efficacy of Intravenous Administration of Human Albumin Versus Saline Solution in Patients With descompénsate Cirrhosis Grade 1B or Higher Renal Failure
Acronym: LIVER-AKI
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Principal Investigator, Anna Cruceta, Clinical Research Manager, Fundacion Clinic per a la Recerca Biomédica
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LIVER-AKI
Record Dates: First submitted 2025-11-14; First posted 2025-12-08 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Decompensated Cirrhosis; AKI - Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This is a phase IV, unicentric, open-label, randomized clinical trial, low interventional level
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Human Albumin (No Intervention): Intravenous Human Albumin 20% (20 g/100 ml), at a dose of 1 g per kg body weight with a maximum of 100 g per day, during 48 hours.
- Saline solution (Experimental): Saline solution (NaCl 0.9%) 500 ml every 24 hours, administered during 48 hours
  Interventions: Drug: Saline solution (NaCl 0.9%)

INTERVENTIONS:
Drug: Saline solution (NaCl 0.9%) — Saline solution (NaCl 0.9%) 500 ml every 24 hours, administered during 48 hours.
  Arms: Saline solution

SUMMARY:
This is a phase IV, unicentric, open-label. Patients eligible for this study will be patients with AKI 1B or greater and decompensated cirrhosis from the hospital participating in the study

DETAILED DESCRIPTION:
This is a phase IV, unicentric, open-label, randomized clinical trial to evaluate the efficacy of intravenous human albumin administration versus saline solution (NaCl 0.9%) in patients with decompensated cirrhosis and AKI 1B or grater.

Patients will be randomized to receive (1:1):

1. Intravenous Human Albumin 20% (20 g/100 ml), at a dose of 1 g per kg body weight with a maximum of 100 g per day, during 48 hours.
2. Saline solution (NaCl 0.9%) 500 ml every 24 hours, administered during 48 hours. Patients will be followed up for 28 days since the administration of the treatment (at baseline visit).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. Cirrhosis defined by standard clinical criteria, ultrasonographic findings and/or histology. (Cirrhosis of any etiology may be included).
3. Patients with AKI 1B or greater, defined according to EASL guidelines (EASL. J Hepatol 2018).
4. Women of child-bearing potential* must have a negative pregnancy test in serum before the inclusion in the study and agree to use highly effective contraceptive methods during the study. Highly effective contraceptive methods will include: intrauterine device, bilateral tubal occlusion, vasectomized partner and sexual abstinence** (only if refraining from heterosexual intercourse during the period of twelve months). Hormonal contraceptive methods will be avoided due to the risk of adverse events and impairment of liver function

Exclusion Criteria:

1. Time since AKI diagnosis > 24 hours.
2. Patients with AKI due to pure hypovolemia. According to guidelines, these patients should receive crystalloid solutions (i.e. NaCl 0.9%) and will be excluded from the study. Fluid losses will be specifically assessed by an accurate anamnesis and physical examination. If patient's diuretic treatment has been increased recently (within prior 2 weeks), or the patient had diarrhea before admission, patient will be considered that the AKI phenotype is pre-renal and will be excluded from the analysis. Patients will be excluded when clear evidence of hypovolemia is present, based on clinical history (e.g, recent fluid losses, diuretic escalation, diarrhea) and corroborating physical findings (e.g, dry mucous membranes, reduced skin turgor, sunken eyes, or low jugular venous pressure)
3. Patients with AKI due to gastrointestinal bleeding with AKI 1B or greater, and hemoglobin < 7.0 g/dL. These patients can be included after 48 hours without rebleeding and Hb ≥ 8.0 g/dL, and still present AKI 1B or greater.
4. Patients who had already received albumin at the time of inclusion/exclusion criteria assessment.
5. Patients with Chronic kidney disease grade 3a or higher, defined as glomerular filtration rate <60ml/min for three months and markers of kidney damage (one or more): Albuminuria (Albumin excretion rate > 30 mg/24h; Albumin-to-creatinine ratio > 30 mg/g), Urine sediment abnormalities, Electrolyte and other abnormalities due to tubular disorders, Abnormalities detected by histology or Structural abnormalities detected by imaging.
6. Patients under renal replacement therapy, or with urgent criteria of RRT.
7. Patients with hepatocellular carcinoma beyond Milan criteria.
8. Patients with severe extrahepatic comorbidities, including congestive heart failure New York Heart Association Grade III/IV, chronic obstructive pulmonary disease Global Initiative for Chronic Obstructive Lung Disease group 2 or higher.
9. Previous liver and/or kidney transplantation.
10. Patients with current extra hepatic malignancies including solid tumors and hematologic disorders.
11. Patients included in other clinical trials in the month before inclusion.
12. Patients with mental incapacity, language barrier, bad social support or any other reason considered by the investigator precluding adequate understanding, cooperation or compliance in the study.
13. Refusal to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
probability of AKI resolution among patients with decompensated cirrhosis and AKI 1B or greater acute kidney injury (AKI) clinical efficacy of HA versus saline (NaCl 0.9%) administration in patients will be evaluated, | at any time during the study (all visits: screenning, basal , day 1, day2, day 5, day 7, day 15, and day 28)
  defining AKI resolution as the proportion of patients with a decrease in serum creatinine levels < 0.3 mg/dL with respect to baseline serum creatinine, without the need for TRT.

SECONDARY OUTCOMES:
Survival rate patients | at 28 days (visit 6)
  Survival rate patients at 28 days, considering liver transplantation as a competitive risk event.
AKI improvement | basal visit , day 1, day2, day 5, day 7, day 15, and day 28)
  defined as the proportion of patients who decrease at least 1 grade of AKI classification (from 3 to 2, from 2 to 1B, and from 1B to 1A or recovery), without the need for RRT.
Proportion of patients requiring RRT In both groups | basal visit , day 1, day2, day 5, day 7, day 15, and day 28)
  Proportion of patients requiring RRT In both groups (renal replacemtent theraphy)
Changes from baseline in systemic inflammatory response, evaluated by measurement in a large array of plasma cytokine levels (IL-6, IL8, IL-10, IL-1β) | basal visit , day 1, day2, day 5, day 7, day 15, and day 28)
  picograms per mililiter (pg/mL)
Changes from baseline in systemic inflammatory response, evaluated by measurement in TNFα, | basal visit , day 1, day2, day 5, day 7, day 15, and day 28)
  picograms per mililiter (pg/mL)
Changes from baseline inG-CSF | basal visit , day 1, day2, day 5, day 7, day 15, and day 28)
  micrograms per kilogram of body weight (mcg/kg)
Changes from baseline in systemic hemodynamics and vasoactive hormones: plasma copeptin | basal visit , day 1, day2, day 5, day 7, day 15, and day 28),
  ypically range from 1 to 13 pmol/L
Changes from baseline in systemic hemodynamics and vasoactive hormones: plasma renin concentration | basal visit , day 1, day2, day 5, day 7, day 15, and day 28)
  ng/mL/hr (nanograms per milliliter per hour)
Changes in echocardiographic parameters (E/E', ITV, among others) at visit 1, 2, 7 and 28. | basal visit , day 1, day2, day 7, day, and day 28)
  (E/E', ITV)
Proportion of patients and severity of treatment-related adverse events during the study period | screening visit,basal visit , day 1, day2, day 5, day 7, day 15, and day 28)
  number and description SAEs and SUSARs

IPD SHARING:
Plan to Share IPD: No